CLINICAL TRIAL: NCT01143324
Title: A Prospective, Multicenter Observational Study on MAST™ (Minimal Access Spinal Technologies) Fusion Procedures for the Treatment of the Degenerative Lumbar Spine (MASTERS-D)
Brief Title: A Prospective, Multicenter Observational Study on MAST™ (Minimal Access Spinal Technologies) Fusion Procedures for the Treatment of the Degenerative Lumbar Spine
Acronym: MASTERS-D
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: MASTERS-D Study
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2016-01

CONDITIONS: Degenerative Lumbar Spine Causing Back and/or Leg Pain; Lumbar Spine Degeneration
Keywords: Single or double level instrumented fusion; Degenerative lumbar spine; PLIF; TLIF; MAST procedure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MAST™ procedure
  Interventions: Device: MAST™ procedure

INTERVENTIONS:
Device: MAST™ procedure — Single or double level instrumented fusion receiving the CD Horizon® Spinal System using PLIF or TLIF techniques via a MAST™ procedure.

SUMMARY:
The aim of the study is to observe and document surgical practice and evaluate patients' outcomes following a MAST™ single or double level instrumented fusion procedure using PLIF (Posterior Lumbar Interbody Fusion) or TLIF (Transforaminal Lumbar Interbody Fusion) techniques for the treatment of the degenerative lumbar spine in a "real-world" patient population.

DETAILED DESCRIPTION:
Instrumented lumbar fusion is usually done through an open procedure which involves an excessive intraoperative dissection and retraction of the paraspinal musculature leading, in a short term basis, to a prolonged recovery time from the surgery. This open approach is frequently associated with significant blood loss and need of transfusion, produces the majority of the perioperative pain, increases hospital stay and the chances of infection and delays the return to normal activities and to work. In a long term basis, the open procedure leads to denervation, atrophy and loss of the muscles independent function, resulting in an increased risk of "fusion disease", a term that has been coined to describe its occurrence.

The minimally invasive spinal surgery was developed as a potential solution to the above-mentioned problems by reducing the amount of iatrogenic soft tissue injury while reaching the same traditional goals of the open procedures. Besides minimizing the long-term effects of exposure-related muscle injury, minimally invasive lumbar fusion techniques hold the promise of immediate short-term advantages. Patients undergoing minimally invasive procedures are reported to recover earlier from the surgery. Shorter time to first ambulation, less pain medication consumption, less blood loss, less required transfusion, shorter hospital stay and earlier return to work are generally associated with the minimally invasive procedure as compared to the standard open surgeries. The minimally invasive access requires a surgical corridor targeted on the disease which is accomplished by using a series of tubular muscle dilators allowing a clear intraoperative visualization to perform these procedures together with the parallel use of image guided percutaneous insertion of pedicle screws and instrumentation.

The purpose of this study is to observe and document surgical practice and evaluate patients' outcomes following a MAST™ single or double level instrumented fusion procedure using PLIF or TLIF techniques for the treatment of the degenerative lumbar spine in a "real-world" patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years of age (or minimum age as required by local regulations).
* Patient has indication for a single or double level instrumented lumbar fusion for the treatment of the degenerative lumbar spine.
* Patient agrees to participate in the study and is able to sign the Data Release Form/Informed Consent.
* The procedure planned for the patient complies with the labeling of the Devices that may be used in the surgical procedure as described in the section B.2 Device Information.
* Patient is planned to be submitted to the fusion procedure using PLIF or TLIF techniques and to receive a CD HORIZON® Spinal System via a MAST™ approach.
* The patient is willing and is able to cooperate with study procedures and required follow-up visits.

Exclusion Criteria:

* Patient that has already undergone an open lumbar spine surgery other than microdiscectomy.
* Indications for the procedure other than degenerative spine disease like Osteoporotic vertebral fractures, Spine trauma fractures and Spine tumor.

In order to reduce as much as possible bias in this observational study, the study centers should propose the study to all consecutive individuals who meet these in and exclusion criteria to participate in the study in order to comply with the 'real world' population concept. This observational study does not require any specific test or procedure that falls outside a standard surgical procedure and patient follow-up as routinely done in the hospital. Some data was collected only for centers that applied such procedures as standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population comprises individuals that have an indication for a single or double level instrumented lumbar fusion for the treatment of the degenerative lumbar spine causing back and/or leg pain.
  Patients enrolled in this study will receive a single or double level instrumented fusion using PLIF or TLIF techniques via a MAST™ procedure.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Franke, PD Dr., Principal Investigator — Klinik für Wirbelsäulenchirurgie; Dortmund
Locations (19):
- Klinikum Amstetten, Amstetten, Austria
- OLV Ziekenhuis, Aalst, Belgium
- Spine, Sports Medicine and Orthopedic Surgery, Saint John, New Brunswick, Canada
- Karvinska Hornicka Nemocnice, Fryštát, Czechia
- Germany (4):
  - Klinikum Kulmbach, Kulmbach, Bavaria
  - Marienhaus Klinikum, Bendorf
  - Neurochirurgische Universitatsklinik, Freiburg im Breisgau
  - Universitätsklinikum Magdeburg, Magdeburg
- Mediterraneo, Glyfada, Greece
- The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Instituto Ortopedici Rizzoli, Bologna
  - Fatebenefratelli Hospital, Milan
- Netherlands (2):
  - Bergman Clinics, Naarden
  - Franciscus Ziekenhuis Roosendaal, Roosendaal
- University Clinical Center, Gdansk, Poland
- Hospital San Joao, Porto, Portugal
- Ustredna Vojenska Nemocnica SNP, Ružomberok, Slovakia
- Hospital Clinic De Barcelona, Barcelona, Spain
- Guys & St; Thomas NHS Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 255 patients were enrolled. Three patients were not submitted to a minimally invasive MAST fusion procedure and therefore excluded from further analysis. Number of participants started in the participant flow is 252.
Groups:
- MAST™ Procedure: Single Arm Study with MAST™ procedure: Single or double level instrumented fusion receiving the CD Horizon® Spinal System using PLIF or TLIF techniques via a MAST™ procedure.
Period: Overall Study
Arm/Group | MAST™ Procedure
Started | 252
Completed | 233
Not Completed | 19
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 4
Not completed — Explant of the device | 4

BASELINE CHARACTERISTICS:
Population: The original CIP planned the enrollment of approximately 200 patients (min 150 and max 250 pts). In total 255 patients were enrolled. Three patients were not submitted to a minimally invasive MAST fusion procedure and therefore excluded from further analysis. The total MAST population analysed at baseline consists of 252 patients.
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 110
Region of Enrollment [Number; unit: Participants] — In total, 255 patients were enrolled, from which 3 patients were not submitted to a minimally invasive MAST fusion and therefore 252 patients were treated and analyzed.
  Participants
    Portugal | 10
    Slovakia | 7
    Greece | 1
    Spain | 4
    Austria | 25
    Israel | 8
    Italy | 16
    United Kingdom | 11
    Czechia | 40
    Canada | 14
    Belgium | 15
    Poland | 4
    Germany | 81
    Netherlands | 16

OUTCOME MEASURES:

1. Primary Outcome: Time From Surgery to First Ambulation.
Description: The primary objective of the study is to access the short term recovery (from surgery to hospital discharge) since the minimally invasive lumbar fusion techniques are expected to be associated with immediate short-term benefits. Patients undergoing minimally invasive procedures are reported to recover earlier from surgery particularly with a shorter time to first ambulation and shorter discharge as compared to the standard open procedures.
  Outcome measure timeframe for time from surgery to first ambulation is assessed up to hospital discharge as pts are all ambulated before discharge from the hospital.
Time Frame: From date of Surgery to date of First ambulation, assessed up to hospital discharge.
Measure: Mean (Standard Deviation); unit: Days from surgery to first ambulation
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Days from surgery to first ambulation | 1.3 (0.5)
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Mean = 1.3, 95% CI 2-sided [1.2 to 1.3], Standard Deviation 0.5

2. Secondary Outcome: Back Pain Intensity Visual Analog Scale (VAS) Score as Compared to Baseline.
Description: Relief of Back Pain intensity at 12 months compared to the baseline using the Back Pain Intensity Score assessed on a 10 cm Visual Analog Scale (VAS).
  The endpoint is the difference between baseline and 12 months of the patient's back-pain intensity score on a Visual Analogue Scale (VAS). A standardized visual analogue scale (0cm-10cm; with 0cm meaning 'no pain' and 10cm meaning 'worst possible pain') was used. Large values of the VAS score represent large degree of pain. Large (negative) change in VAS score (12 months - baseline) represents large relief of pain.
Time Frame: Baseline, 12 months
Population: The number of analyzed at 12 months only included subjects who had available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Units on a scale
  Pre-operative (N=252) | 6.2 (2.3)
  12 Months (N=226): number analyzed (Participants) | 226
  12 Months (N=226) | 2.9 (2.5)
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Difference from pre-op mean = -3.3, 95% CI 2-sided [-3.6 to -2.9]

3. Secondary Outcome: Leg Pain Intensity VAS Score as Compared to Baseline
Description: Leg pain intensity (using VAS intensity score) as compared to baseline. Relief of Leg Pain intensity at 12 months compared to the baseline using the Back Pain Intensity Score assessed on a 10 cm Visual Analog Scale (VAS).
  The endpoint is the difference between baseline and 12 months of the patient's leg-pain intensity score on a Visual Analogue Scale (VAS). A standardized visual analogue scale (0cm-10cm; with 0cm meaning 'no pain' and 10cm meaning 'worst possible pain') was used. Large values of the VAS score represent large degree of pain. Large (negative) change in VAS score (12 months - baseline) represents large relief of pain.
Time Frame: Baseline, 12 months
Population: The number of analyzed at 12 months only included subjects who had available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Units on a scale
  Baseline (N=252) | 5.9 (2.8)
  12 months (N=226): number analyzed (Participants) | 226
  12 months (N=226) | 2.2 (2.6)
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Difference from pre-op mean = -3.8, 95% CI 2-sided [-4.2 to -3.3]

4. Secondary Outcome: EQ-5D Questionnaire (When it is a Routine Practice) as Compared to Baseline.
Description: EQ-5D questionnaire as compared to baseline measurement. EQ-5D Index was calculated based on answers provided in the questionnaire. Applicable to a wide range of health conditions and treatments, the EQ-5D provides a simple descriptive profile and a single index value for health status. The EQ-5D-3L consists of the EQ-5D-3L descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking in the box against the most appropriate statement in each of the 5 dimensions. EQ VAS records the respondent's self-rated health on a vertical 20 cm VAS where the endpoints are labelled 'Best imaginable health state' at the top and 'Worst imaginable health state' at the bottom, having numeric values of 100 and 0 respectively.
Time Frame: Baseline, 12 months
Population: The number of analyzed at 12 months only included subjects who had available data.
Measure: Mean (Standard Deviation); unit: Units on a scale / Index
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 204
Units on a scale / Index
  Baseline (N=204) | 0.34 (0.32)
  12 Months (N=182): number analyzed (Participants) | 182
  12 Months (N=182) | 0.71 (0.28)
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Difference from pre-op mean = 0.35, 95% CI 2-sided [0.30 to 0.41]

5. Secondary Outcome: Fusion Rate as Assessed by CT Scan or X-Rays, in Those Sites Where This Assessment is Standard of Care.
Description: Fusion rate as assessed by the CT Scan or X-Rays, in those sites where this assessment is standard of care.
Time Frame: 12 months
Population: One hundred and thirty one-level patients (=130 LEVELS) and 24 two-level patients (=48 LEVELS) were assessed for fusion at 12 months per CIP defined criteria.
Measure: Number; unit: Fused levels
Units Other Than Participants: Number of levels assessed
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 154
Number analyzed (Number of levels assessed) | 178
Fused levels
  One level fusion (levels n=130): number analyzed (Number of levels assessed) | 130
  One level fusion (levels n=130) | 118
  Two level fusion (levels n=48): number analyzed (Number of levels assessed) | 48
  Two level fusion (levels n=48) | 43

6. Secondary Outcome: Number of Patients Who Utilized Rehabilitation Programs
Description: The number of patients who utilized rehabilitation programs was documented (when required).
Time Frame: From 6-12 months after the day of surgery
Measure: Number; unit: participants
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
participants | 61
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Percentage = 27.0 — 61/226 patients underwent a rehabilitation programs between 6 and 12 months follow up visit, making it 27.0 % of the total

7. Secondary Outcome: Proportion of Patients Needing a Second Intervention at the Treated Level(s) (Reoperation Rates).
Description: Proportion of the patients needing a second intervention at the treated level(s) (reoperation rates).
Time Frame: From baseline until 12 months
Measure: Number; unit: Participants
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Participants | 3
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Percentage = 1.2 — The rate of additional lumbar spinal surgeries at treated level was 1.2% (3/252) patients

8. Secondary Outcome: Proportion of Patients Needing Intervention at Adjacent Level(s).
Description: Proportion of the patients needing intervention at adjacent level(s).
Time Frame: From Baseline until 12 months
Measure: Number; unit: Participants
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Participants | 4
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Percentage = 1.6 — The rate of additional lumbar spinal surgeries at the same level was 1.6% (4/252) patients

9. Secondary Outcome: Document Change in Pain Medication Consumption Over Time as Compared With Baseline. Baseline.
Description: Document the change in pain medication consumption one year after surgery , as compared with baseline. The endpoint is the number of participants taking pain medication at baseline and number of participants taking pain medication in the week before the 12 months follow up visit.
Time Frame: Baseline, 12 months
Population: The number of analyzed at 12 months only included subjects who had available data.
Measure: Number; unit: Participants
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Participants
  Participants taking medication at baseline N=252 | 185
  Participants taking medication at 12 months N=233: number analyzed (Participants) | 233
  Participants taking medication at 12 months N=233 | 107
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Percentage at 12 months = 47.6

10. Secondary Outcome: Document Adverse Events Occurrence Throughout the Study.
Description: Document the Adverse Events occurrence throughout the study. All adverse events have been included regardless visit windowing.
Time Frame: From Baseline until 12 months
Measure: Number; unit: Number of reported adverse events
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Number of reported adverse events | 125

11. Secondary Outcome: ODI Difference 12 Months After the Surgery as Compared to Baseline.
Description: Oswestry Disability Index (ODI) 12 months after the surgery as compared to baseline. The Oswestry Disability Index (ODI) derives from the Oswestry Low Back Pain Questionnaire, it is used to measure disability for low back pain. The index is scored from 0 to 100; 0 meaning 'no disability' and 100 meaning 'maximum disability'.
Time Frame: Baseline, 12 months
Population: The number of analyzed at 12 months only included subjects who had available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 251
Units on a scale
  Baseline (N=251) | 45.5 (15.4)
  12 Month (N=226): number analyzed (Participants) | 226
  12 Month (N=226) | 22.4 (18.8)
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Difference from pre-op mean = -23.0, 95% CI 2-sided [-25.5 to -20.5]

12. Secondary Outcome: Number of Patients That Returned to Work 12months After the Surgery.
Description: Document number of participants that returned to work 12 months after surgery.
Time Frame: 12 months after the surgery
Population: The analyzed subjects at 12 months only included the subjects who had available data.
Measure: Number; unit: Participants currently working
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Participants currently working
  Number of participants working at baseline(N=252) | 79
  Number of participants working at 12 months (N=227: number analyzed (Participants) | 227
  Number of participants working at 12 months (N=227 | 97
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Percentage = 42.7

13. Primary Outcome: Time to Surgery Recovery Day.
Description: The primary objective of the study is to access the short term recovery (from surgery to discharge) since the minimally invasive lumbar fusion techniques are expected to be associated with immediate short-term benefits. Patients undergoing minimally invasive procedures are reported to recover earlier from surgery particularly with a shorter time to first ambulation and shorter discharge as compared to the standard open procedures.
  Surgery recovery day is defined as the day when patients fulfils following criteria : patient no longer needs intravenous infusion of analgesic drugs, there are no surgery related complications (AEs) impending discharge of patient, patient no longer needs nursing care. The objective of the surgery recovery day assessment is to collect the day when the patient could be discharged based on his actual clinical condition because the effective day of discharge may be prolonged by factors other than the patient's clinical recovery such as social factors.
Time Frame: From date of surgery until date of surgery recovery day assessed up to hospital discharge.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MAST™ Procedure
Number analyzed (Participants) | 252
Days | 3.2 (2.0)
Statistical Analysis 1: Comparison: MAST™ Procedure; Test type: Superiority or Other; Mean = 3.2, 95% CI [2.9 to 3.4], Standard Deviation 2.0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | MAST™ Procedure
Serious Adverse Events (participants affected / at risk) | 20/252
Other Adverse Events (participants affected / at risk) | 66/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAST™ Procedure (N=252)
Hypotension (Vascular disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Circulatory collapse (Vascular disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Bladder neck suspension (Surgical and medical procedures) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Spinal haematoma (Nervous system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAST™ Procedure (N=252)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (31)
Cataract (Eye disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Dural tear (Injury, poisoning and procedural complications) | 4 (4)
Pyrexia (General disorders) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoesthesia (Nervous system disorders) | 3 (3)
Implant site effusion (General disorders) | 2 (2)
Incision site abscess (Infections and infestations) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (30)
Lumbar radiculopathy (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study include the lack of a direct comparison of outcomes of minimally invasive surgery and open surgery, since it was designed as an observational trial and not designed as a randomized controlled trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential Disclosure Agreements were signed by all investigators. The information had to be kept confidential and investigators agreed not to disclose information to any third party.